CLINICAL TRIAL: NCT05191186
Title: Documentation of Efficacy of Intralymphatic Allergen Immunotherapy in a Phase III Randomized, Parallel Group Placebo Controlled Double Blind Multisite Field Trial
Brief Title: Documentation of Efficacy of Intralymphatic Allergen Immunotherapy
Acronym: ILITNU
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: University of Aarhus (Other); University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Johannes Martin Schmid, Consultant, MD, PhD, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020-001060-28
Record Dates: First submitted 2021-12-27; First posted 2022-01-13 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Allergic Rhinitis Due to Grass Pollen; Allergic Conjunctivitis of Both Eyes; Allergic Asthma
Keywords: Allergen immunotherapy; Allergic rhinoconjunctivitis; grass pollen allergy; intralymphatic immunotherapy; ILIT.NU
MeSH Terms: interventions — Immunotherapy

STUDY DESIGN:
Intervention Model Description: parallel group, double blind placebo controlled multi site
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study is run in a double-blind design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- grass pollen extract treatment (Active Comparator): participants receive 3 injections with Alutard phleum pratense, ALK, grass pollen extract
  Interventions: Drug: Grass pollen extract - Alutard Phleum pratense, ALK
- Placebo (Placebo Comparator): Participants receive 3 injections with saline (NaCl 0.9%)
  Interventions: Drug: Grass pollen extract - Alutard Phleum pratense, ALK

INTERVENTIONS:
Drug: Grass pollen extract - Alutard Phleum pratense, ALK — injection in lymph node
  Other Names: immunotherapy

SUMMARY:
Investigation of the clinical efficacy of 3 intralymphatic injections with grass pollen extract into inguinal lymph nodes on combined symptom-medication scores during grass pollen season in grass pollen allergic patients compared to placebo

DETAILED DESCRIPTION:
A double-blind, parallel group, placebo controlled multi-site trial of the clinical efficacy of 3 intralymphatic injections with a low dose of grass pollen extract into inguinal lymph nodes in grass pollen allergic subjects.

Primary endpoint is the difference in combined symptom and medication score during grass pollen seasons following treatment compared with patients receiving placebo.

Injections are giving ultrasound-guided with at least 4 weeks intervals.

To increase trial retention, two studies within the trial are conducted: a feasibility study assessing the acceptability and feasibility of a digital intervention and its evaluation design. Outcomes include participant and stakeholder acceptability, reach, mechanisms of change to improve trial retention, utilization, unintended effects, software functionality, recruitment and retention rates, questionnaire suitability, randomization feasibility, power for a future definitive trial, and initial efficacy signals. Additionally, an evaluation study assesses the efficacy of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* moderate-severe grass pollen allergic rhinoconjunctivitis
* positive skin prick test for grass pollen extract

Exclusion Criteria:

* significant mugwort allergy
* previous AIT for grass pollen allergy
* uncontrolled non-allergic upper airways disease
* uncontrolled asthma
* planned depot steroid injections during season
* uncontrolled autoimmune diseases
* active malignancies
* uncontrolled other severe condition, including psychiatric diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Combined symptom and medication score, cSMS | 2 years
  daily combined symptom and medication scores during grass pollen seasons in 2022 and 2023 as compared to placebo.
  cSMS is a combined score of a symptom score, 0-3, where 0 indicates no symptoms and 3 indicates severe symptoms and meddication score 0-3 according to the us of reliever medication: 0: no medication, 1: antihistamine use, 2: local steroid use, 3: systemic steroid use.
  This results in a score ranging from 0 (no symptoms, no need for medications) to 6 (severe symptoms and need for maximum reliever medication

SECONDARY OUTCOMES:
side-effects | 3 months
  occurence of side-effects as compared to placebo
correlation of CSMS to pollen count | 2 years
  correlate cSMS to daily pollen counts
combined symptom and medication score, cSMS | 2 years
  change in the combined symptom and medication score from baseline
Rhinitis related quality of life, RQLQ | 2 years
  changes on rhinitis related quality of life
Airwave oscillometry system(AOS), asthma | 2 years
  Influence of ILIT on resistance in the lower airways measured by AOS

CONTACTS AND LOCATIONS:
Overall Officials: Johannes M Schmid, MD PhD, Principal Investigator — Aarhus University Hospital/Aarhus University
Locations (2):
- Aarhus University Hospital, Aarhus, Central Region, Denmark
- Linkoeping University Hospital, Linköping, Oestergotland, Sweden

IPD SHARING:
Plan to Share IPD: No
We will publish data

REFERENCES:
- [Derived] Petersen AP, Schmid JM, Hoffmann HJ, Finderup J. Acceptability and feasibility of a need-supportive intervention to increase trial retention: a randomised feasibility study within a randomised controlled allergy trial in Denmark. BMJ Open. 2025 Sep 14;15(9):e101046. doi: 10.1136/bmjopen-2025-101046. PMID 40953876
- See also: project homepage — http://ILIT.NU